CLINICAL TRIAL: NCT05266105
Title: A Phase 1 Dose Escalation and Expansion Open-label, Multicenter, Study of OP-1250 in Combination With the CDK4/6 Inhibitor Palbociclib in Adult Subjects With Advanced or Metastatic HR-positive, HER2-negative Breast Cancer
Brief Title: A Phase 1 Study of Oral OP-1250 in Combination With Palbociclib in HR+/HER2- Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-1250-002
Record Dates: First submitted 2022-02-11; First posted 2022-03-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Escalation (Experimental): This portion of the study will evaluate the safety and pharmacology of a range of OP-1250 doses administered daily with Palbociclib in subjects with advanced and/or metastatic hormone receptor (HR)-positive, HER2-negative breast cancer
  Interventions: Drug: Palazestrant; Drug: Palbociclib
- Dose Expansion (Experimental): This portion of the study further explores the clinical activity, safety and pharmacology of OP-1250 in combination with Palbociclib and estimates preliminary data of anti-tumor efficacy
  Interventions: Drug: Palazestrant; Drug: Palbociclib

INTERVENTIONS:
Drug: Palazestrant — Complete Estrogen Receptor Antagonist
  Other Names: OP-1250
Drug: Palbociclib — Palbociclib is an approved CDK 4/6 Inhibitor drug
  Other Names: Ibrance®️

SUMMARY:
This is an open-label, Phase 1b dose escalation and expansion study to determine the maximum tolerated dose (MTD) of OP-1250 in combination with palbociclib (Ibrance®️, Pfizer Inc.). Purpose of study is to evaluate the safety and pharmacokinetic (PK) profile, and estimate the preliminary anti-tumor activity of the combination in adult subjects with hormone receptor-positive (ER+ / HER2-) advanced or metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed and evaluable locally advanced or metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Must not have received prior oral endocrine or targeted therapy ≤ 2 weeks prior to first dose
* Must not have received prior chemotherapy, antibody therapy, or investigational therapy ≤ 4 weeks prior to the first dose
* Prior radiotherapy must have been completed 2 weeks prior to first dose
* Adequate safety laboratory tests
* Willingness to use effective contraception

Exclusion Criteria:

* Gastrointestinal disease
* Significant hepatic disease
* Significant cardiovascular disease
* Significant ECG abnormalities
* History of pulmonary embolism or high risk of thrombosis
* Known HIV infection
* Active infection (requiring antimicrobial therapy)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | From Cycle 1 Day 1 through C1 Day 28
Characterization and Incidence in Adverse Events and Serious Adverse Events | From initial inform consent date through 30 days post last dose
Plasma levels of OP-1250 and Palbociclib | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sue Johnson, Study Director — Olema Pharmaceuticals, Inc.
Locations (8):
- Australia (8):
  - Clinical Trial Site, Waratah, New South Wales
  - Clinical Trial Site, Westmead, New South Wales
  - Clinical Trial Site, South Brisbane, Queensland
  - Clinical Trial Site, Southport, Queensland
  - Clinical Trial Site, Clayton, Victoria
  - Clinical Trial Site, Frankston, Victoria
  - Clinical Trial Site, Geelong, Victoria
  - Clinical Trial Site, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No